CLINICAL TRIAL: NCT05502042
Title: Case Managers and Peer Support Groups (CAMPS) for Prophylaxis Adherence in Rheumatic Heart Disease
Brief Title: Case Management and Peer Support Groups for Prophylaxis Adherence in Rheumatic Heart Disease
Acronym: CAMPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Uganda Heart Institute (Other)
Responsible Party: Principal Investigator, Sarah deLoizaga Carney, Instructor, Pediatrics, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-0789
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Rheumatic Heart Disease
Keywords: adherence; clinical trial; community intervention
MeSH Terms: conditions — Rheumatic Heart Disease | interventions — Case Managers

STUDY DESIGN:
Intervention Model Description: Case Managers and Peer Support Groups (CAMPS) will be a pragmatic randomized trial of two support strategies for rheumatic heart disease secondary antibiotic prophylaxis, integrated into routine care.
Who Masked: Outcomes Assessor
Masking Description: Our primary outcome, adherence to SAP, will be abstracted from copies of final Uganda Ministry of Health SAP booklets by a team member blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Referral to a health facility (HC III, IV, or district hospital) that provide secondary antibiotic prophylaxis (every-28-day intramuscular benzathine benzylpenicillin G, BPG), receipt of a Ministry of Health secondary prophylaxis adherence booklet, and education for patient and family about the importance of SAP.
- Peer Group + Case Manager (Experimental): Usual care + an assigned village health team member to provide weekly short message (SMS) (weeks 1-3) and phone (week 4) support for attendance of SAP visits and a VHT (village health team member) led peer support group held at the assigned SAP clinic of participants, that includes games/peer support/education.
  Interventions: Behavioral: Case Manager and Peer Support Group

INTERVENTIONS:
Behavioral: Case Manager and Peer Support Group — Assignment of a Village health team member to provide support to the family through SMS messages (weeks 1-3) and phone call (week 4), as well as home visits as needed if no contacts are reached. These contacts are intended to provide encouragement and education to participants and families to encourage SAP and peer group attendance. Peer groups will have simple play and support activities, led by the village health team member, to improve the experience of SAP for the participating children.
  Arms: Peer Group + Case Manager

SUMMARY:
The objective of CAMPS is to test and evaluate scalable models of secondary antibiotic adherence support for children newly diagnosed with rheumatic heart disease.

Aim 1: Determine 1-year BPG adherence rates of children newly diagnosed with latent RHD in Uganda randomized to two support strategies: (1) Usual care (Arm 1) (2) peer group + case manager strategy (Arm 2).

Aim 2: Explore patient reported outcomes including treatment satisfaction, patient health-related quality of life, and care giver quality of life, in relation to support strategy and adherence.

DETAILED DESCRIPTION:
While significant strides have been made in echo screening for early detection of RHD and establishment of RHD registries, these efforts are diluted by poor adherence to secondary antibiotic prophylaxis (SAP). In a systematic review by Kevat et al which included 20 global programs, only 20% were able to maintain patients on at least 80% adherence (the minimum acceptable level). Other studies demonstrate similar findings, with adherence ranging from as low as 20% up to 75%. These studies demonstrate that non-adherence undermines most global SAP programs.

Despite low adherence to RHD secondary prophylaxis globally, studies have demonstrated that ideal RHD SAP adherence can be achieved, but within the confines of strict trial conditions (GOAL Trial). Currently, there is a dearth of research into pragmatic, scalable approaches to improve RHD SAP adherence. In their systematic review of effectiveness and integration of RHD prevention and control programs, Abrams et. al. advise that prevention and treatment programs should be integrated into general health systems and strengthen local systems. Case Managers and Peer Support Groups (CAMPS) will be a pragmatic randomized trial of two support strategies for rheumatic heart disease secondary antibiotic prophylaxis, integrated into routine care. Hence, CAMPS will address the gap that exists between ideal adherence achieved within the confines of a strict research trial and practical and scalable solutions that can be translated to real-world settings.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 5-17
2. New diagnosis of latent rheumatic heart disease (RHD) as determined through school screening -

Exclusion Criteria:

1. Medical contraindication to SAP (bleeding risk, allergy)
2. Co-morbid conditions that have already resulted in prescription of SAP (typically HIV, sickle cell disease, renal disease)

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 209 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Secondary Prophylaxis Adherence | 12 months
  Continuous adherence to intramuscular Benzathine penicillin, as determined by days of coverage (each injection = 28 days of coverage)

SECONDARY OUTCOMES:
Treatment satisfaction | 6 months + 12 months
  14-item Abbreviated Treatment Satisfaction Questionnaire (v 1.4)
Patient health-related quality of life | enrollment, 6-months, 12-months
  Pediatric Quality of Life Inventory Version 4.0 Generic Core (PedsQL 4.0) questionnaire
Caregiver health-related quality of life | enrollment, 6-months, 12-months
  Parent/caregiver module of the PedsQL 4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Tororo Health Distric, Tororo, Uganda

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be available to other investigators on reasonable request after publication of the primary results.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of the primary study results (anticipated December 2024)
Access Criteria: Reasonable request for related research

REFERENCES:
- [Derived] de Loizaga S, Pulle J, Atanas O, Alepere J, Nambogo JL, Ndagire E, Kaudha G, Ollberding NJ, Okello E, Rwebembera J, Beaton A. Enhanced support for adherence to rheumatic heart disease prophylaxis for children in the public health system in Uganda (CAMPS): a pragmatic randomised trial. Lancet Glob Health. 2025 Apr;13(4):e707-e715. doi: 10.1016/S2214-109X(24)00527-8. PMID 40155108